CLINICAL TRIAL: NCT06674057
Title: Additional Effects of Kinesio-Taping Along with Conservative Physical Therapy on Upper Limb Function, Range of Motion and Spasticity in the Patients with Subacute Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/42
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Subacute Stroke; Upper Limb; Range of Motion; Spasticity; CVA (Cerebrovascular Accident); KINESIOTAPING; Stroke; Function
Keywords: Stroke.; subacute stroke; kinesio taping; proprioceptive neuromuscular facilitation; Upper limb function.; range of motion
MeSH Terms: conditions — Muscle Spasticity; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental group (Experimental): It includes participants receiving kinesio taping in addition to conservational physical therapy for subacute stroke patient's upper limb ROM/spasticity/function. for a period of 6 weeks.
  Interventions: Procedure: KinesioTaping
- control group (Active Comparator): It includes participants receiving conservational physical therapy for subacute stroke patient's upper limb ROM/spasticity/function. for a period of 6 weeks.
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: KinesioTaping — The experimental group will receive the following treatment for week 1-3 (3 days on alternate days):
  * Passive and active ROMs 25 repetitions each, 3 times per week.
  * PNF stretching (hold relax) for spastic muscles for 20 repetitions with a 10 second hold and 10 second relaxation of the muscle group 3 times per week.
  * D1 flexion and extension for 20 repetitions 3 times per week.
  * Kinesio tape 3 times per week. (Anchor opposed to effected compartment to provide facilitation and sustained stretch).
  For week 3-6 the treatment will include:
  * Passive and active ROMs 25 repetitions each, 3 times per week.
  * PNF stretching (hold relax) for spastic muscles for 20 repetitions with a 10 second hold and 10 second relaxation of the muscle group 3 times per week.
  * D1 flexion and extension for 20 repetitions 3 times per week.
  * Strengthening affected muscle groups by resistance training, 3 times per week (using a resistance band of mediu
  Arms: experimental group
Procedure: Control — The control group will receive the following treatment for week 1-3 on alternate days:
  * Passive and active ROMs 25 repetitions each, 3 times per week.
  * PNF stretching (hold relax) for spastic muscles for 20 repetitions with a 10 second hold and 10 second relaxation of the muscle group 3 times per week.
  * D1 flexion and extension for 20 repetitions 3 times per week.
  For week 3-6 the treatment will include:
  * Passive and active ROMs 25 repetitions each, 3 times per week.
  * PNF stretching (hold relax) for spastic muscles for 20 repetitions with a 10 second hold and 10 second relaxation of the muscle group 3 times per week.
  * D1 flexion and extension for 20 repetitions 3 times per week.
  * Strengthening affected muscle groups by resistance training, 3 times per week (using a resistance band of medium resistance).
  Arms: control group

SUMMARY:
A randomized control trial will be done on diagnosed stroke patients of subacute stage in Fauji Foundation Hospital Rawalpindi and leading edge physical therapy and rehabilitation clinic.The purpose of the study is to determine Additional Effects of Kinesio-Taping along with conservative Physical Therapy on upper limb function, Range of motion and Spasticity in the patients with Subacute Stroke. The conservational physical therapy includes Passive and active ROMs 25 repetitions each, 3 times per week. PNF stretching (hold relax) for spastic muscles for 20 repetitions with a 10 second hold and 10 second relaxation of the muscle group 3 times per week.

D1 flexion and extension for 20 repetitions 3 times per week. Kinesio tape 3 times per week. (Anchor opposed to effected compartment to provide facilitation and sustained stretch). with srtrngth training included in week 3-6 with a resistance band of medium resistance.

treatment time will be 30 minutes on alternate days for six weeks.

DETAILED DESCRIPTION:
OBJECTIVES:

The objectives of this study are:

1. To determine the additional effects of kinesio taping in combination with physical therapy on ROM of upper limb shoulder, elbow and wrist joint in subacute stroke patients
2. To determine the additional effects of kinesio taping in combination with physical therapy on upper limb spasticity in subacute stroke patients
3. To determine the effects of kinesio taping on upper limb function in subacute stroke patients.

HYPOTHESIS:

Alternate Hypothesis:

There is a statistically significant difference between kinesio taping combined with physical therapy on ROM, spacticity and function of upper limb Shoulder, elbow and wrist joints in patients with subacute stroke compared to conventional physical therapy.

Null Hypothesis:

There is no statistically significant difference between kinesio taping combined with physical therapy on ROM, spacticity and function of upper limb Shoulder, elbow and wrist joints in patients with subacute stroke compared to conventional physical therapy.

Research Design: Experimental study. Randomized Control Trial

Clinical setting: Rehabilitation department, Fauji Foundation Hospital , leading edge physical therapy and rehabilitation islamabad.

Study duration: 6 months.

Selection Criteria:

Inclusion Criteria

* Age group: 40-65 years onwards
* Both males and females
* Patients with history of diagnosed stroke and lie within subacute stage of stroke
* MAS scale score of 1_2

Exclusion Criteria

* Any congenital deformities
* cognitive deficits
* Fractures
* Upper limb surgery

Sampling technique: Convenience sampling

Outcome Measures:

Data will be collected on Demographics and general information Goniometer will be used to assess the range of motion of shoulder, elbow and wrist joint Modified Ashworth scale will be used to determine the level of spasticity in the participants.

Wolf motor function test scale for upper limb will be used to assess upper limb function.

Experimental Group (A) = This group will receive kinesio taping every alternate day for six weeks combined with conservational physical therapy which includes AROMs, PROMs, PNF D1 flexion and extension, resistance raining using resistance band of medium resistane.

and their outcomes will be measured at baseline and at 3rd week and at the end of 6th week treatment.

Control group (B) =this group will not receieve kinesio taping , only conservationall Physical therapy will be given and their outcomes will be observed at the baseline, at third week and then after treatment of 06 weeks.

Data analysis techniques:

The data will be analyzed through SPSS 21 and Data would be analyzed based on the study design chosen that is random control experimental study.

A printed questionnaire will be provided to the participents after obtaining written consent and providing adequate explanation regarding the study, after which the data will be presented in the form of graphs or tables.

Significance of the study:

This study will add data to the literature. Providing evidence-based data and aiding healthcare providers to incorporate kinesio taping as an adjunct intervention.

This study will also provide a feasible and cost-effective treatment to the patient diagnosed with subacute stroke.

Kinesio taping is easy to apply, potentially beneficial treatment options for patients with subacute stroke upper limb dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Age group: 40-65 years onwards
* Both males and females
* Patients with history of diagnosed stroke and lie within subacute stage of stroke
* MAS scale score of 1_2

Exclusion Criteria:

* Any congenital deformities
* cognitive deficits
* Fractures
* Upper limb surgery

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
Spasticity | 6 weeks
  velocity dependant passive resistance to stretch will be assesed using the modified ashworth scale.
Upper limb function | 6 weeks
  Upper limb function will be assessed using the wolf motor function test for upper limb.

SECONDARY OUTCOMES:
Range of motion | 6 weeks
  range of motion of Wrist, Elbow and shoulder joint will be assessed using a goiniometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Thrapy, Islamabad, Pakistan